CLINICAL TRIAL: NCT01552941
Title: Pilot Study of the Safety and Efficacy of Neurostimulation of the Cholinergic Anti-Inflammatory Pathway Using an Active Implantable Vagal Nerve Stimulation Device in Patients With Rheumatoid Arthritis
Brief Title: Safety and Efficacy Vagal Nerve Stimulation in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPM-005
Record Dates: First submitted 2012-03-08; First posted 2012-03-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Vagus Nerve; Vagal Nerve Stimulation; Rheumatoid Arthritis; Implantable Medical Device
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vagal Nerve Stimulation (Experimental)
  Interventions: Device: Cyberonics VNS System

INTERVENTIONS:
Device: Cyberonics VNS System — Active Implantable Electrical Vagal Nerve Stimulator

SUMMARY:
This is a 12 week open label pilot study to determine the efficacy and safety of a surgically implanted, electrically active vagal nerve stimulation device in patients with active rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Adult-onset rheumatoid arthritis of at least six months duration as defined by the 2010 ACR/EULAR classification criteria (Aletaha, 2010)
* Male or female patients, 18-75 years of age, inclusive
* Functional status I, II, or III as classified according to the ACR 1991 revised criteria (Hochberg, 1992)
* Patients must have active disease as defined by at least 4 active tender or swollen joints and CRP above 0.7 mg/dL, despite at least 3 months of treatment with methotrexate at a dose of up to 25 mg orally per week.
* Patients may have been previously treated with TNF antagonists, but must have failed by reason of inadequate safety, intolerance to side effects, or development of antibodies (i.e., secondary failures), and specifically cannot have failed on the basis of primary lack of efficacy
* Study amended to add a second cohort of up to 10 patients who have failed both a TNF antagonist and at least one other biological therapy having a non-TNF antagonist mechanism of action

Exclusion Criteria:

* History of unilateral or bilateral vagotomy
* History of recurrent vaso-vagal syncope episodes
* Known obstructive sleep apnea
* Known history of cardiac rhythm disturbances, atrio-ventricular block of greater than first degree, or cardiac conduction pathway abnormalities other than isolated right bundle branch block or isolated left anterior fascicle block
* Significant pharyngeal dysfunction or swallowing difficulties
* Pre-existing clinically significant vocal cord damage or hoarseness
* Previously implanted electrically active medical devices (e.g., cardiac pacemakers, automatic implantable cardioverter-defibrillators)
* Asthma or chronic obstructive pulmonary disease not controlled by medications, or any other disease causing clinically significant dyspnea at time of screening
* Active peptic ulcer disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in DAS from baseline | 6 weeks

SECONDARY OUTCOMES:
Number of patients with ACR 20 response | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Peter Tak, M.D., Ph.D., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (4):
- Bosnia and Herzegovina (2):
  - Sveučilišna klinička bolnica Mostar, Mostar
  - Klinicki Centar Univerziteta, Reumatologija, Sarajevo
- Sisters of Mercy Clinical Hospital Centre, Zagreb, Croatia
- Academic Medical Center, University of Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koopman FA, Chavan SS, Miljko S, Grazio S, Sokolovic S, Schuurman PR, Mehta AD, Levine YA, Faltys M, Zitnik R, Tracey KJ, Tak PP. Vagus nerve stimulation inhibits cytokine production and attenuates disease severity in rheumatoid arthritis. Proc Natl Acad Sci U S A. 2016 Jul 19;113(29):8284-9. doi: 10.1073/pnas.1605635113. Epub 2016 Jul 5. PMID 27382171